CLINICAL TRIAL: NCT07367828
Title: Feasibility and Validity of Frailty Screening Tools as a Measure of Postoperative Outcomes in Older Patients Undergoing Elective Surgery
Brief Title: Validity of Frailty Screening Tools as a Measure for Postoperative Outcomes
Status: Recruiting | Type: Observational
Sponsor: University of Iceland (Other)
Collaborators: Landspitali University Hospital (Other)
Responsible Party: Principal Investigator, Martin Ingi Sigurdsson, Professor in Anesthesiology and Intensive Care, University of Iceland
Other Study IDs: VRN 25/2024
Record Dates: First submitted 2025-12-12; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Frailty in Adult Surgery; Frailty Syndrome; Elective Surgery
Keywords: Frailty; Postoperative Outcomes; Major elective surgery; Surgical Frailty; Intermediate elective surgery
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Frailty screening cohort: The study will consist of a cohort of surgical patients ≥ 70 years undergoing Intermediate/major elective surgery who present for preoperative assessment at the anesthesia outpatient clinic at Landspitali - The National University Hospital in Iceland.
  Patients who screen positive on the CDT (≤ 2/3 points) and TUG (≥ 11 seconds) will be considered frail. Those who do not screen positive on both of these tests will be part of the control group (non-frail).
  Interventions: Procedure: Intermediate/major elective surgery

INTERVENTIONS:
Procedure: Intermediate/major elective surgery — Any intermediate/major elective surgery at Landspítali -The National University Hospital in Iceland

SUMMARY:
Frailty is a common geriatric syndrome defined as a clinical state of decreased physiologic reserve resulting in increased vulnerability to stressors. It is associated with several unfavorable postoperative complications independent of age such as readmission, length of hospital stay and mortality. To address these concerns, medical societies have acknowledged a need for routine screening to identify elderly patients who are at high risk for major complications before undergoing surgery.

In the absence of a golden standard for frailty assessment, there are multiple assessment tools available. However, the challenge with many frailty tools is that they can be time-consuming, and require expertise and clinical training.This poses a challenge for screening a large elderly population before surgery. Some frailty assessment tools, such as PRISMA7 (The Program of Research to Integrate Services for the Maintenance of Autonomy), timed up and go (TUG) and the clock drawing test (CDT), have been demonstrated to be quick, simple and easy to use with minimal training.

The PRISMA-7 is a frailty screening questionnaire that consists of seven dichotomous items considering age, gender, health problems that affect activities of daily living (ADLs), assistance from others with ADLs, having to count on someone if needed, and the use of mobility aids.

The TUG test is used for assessing fall risk and frailty in older patients. It is measured by the time it takes an individual to stand up from a seated position, walk three meters and return back to a seated position. There is no standard cut-off for TUG, however, a cut-off of > 10 seconds has been used to identify frailty.

Cognitive impairment in older surgical patients may predispose patients to executive dysfunction that many elderly patients experience postoperatively and has shown to be a risk factor for surgical complications. Some studies suggest a strong relationship between cognitive impairment and physical frailty resulting in cognitive frailty when evaluating older adults.The CDT has shown to be a valuable screening tool for cognitive concerns. When administering the CDT, a patient receives instructions to draw a clock. Performing the test requires auditory comprehension, planning, sustained attention, visual-spatial skills and executive skills.

The prevalence of surgical frailty in Iceland has not been researched thoroughly enough to provide an accurate estimate. This is important to reveal the number of senior surgical patients at high risk of adverse postoperative outcomes who could benefit from a preoperative intervention. However, there is a lack of consensus on an optimal frailty assessment to screen patients for identifying frail patients prior to surgery, and more research is needed to evaluate which group of patients would benefit the most from prehabilitation.

The scientific value of this study is to elucidate the extent of frailty risk and its associated postoperative outcomes in older surgical patients undergoing elective surgery. We opt to find a convenient screening routine prior to surgery to identify patients at risk of frailty. Therefore, the study aims to validate three frailty screening methods and to assess a positive screening result as an independent risk factor for adverse postoperative outcomes in a cohort of elderly surgical patients undergoing elective surgery. We hypothesize that elderly patients at risk of frailty have a higher rate of surgical complications than patients not at risk of frailty.

Patients aged ≥ 70 years who undergo elective surgery will be prospectively examined at the Department of Anesthesiology and Critical Care of Landspítali. The screening assessments to be evaluated are the Program of Research to Integrate Services for the Maintenance of Autonomy (PRISMA-7), a combination of Timed Up & Go (TUG), Clock Drawing Test (CDT) and the FRAIL questionnaire, and a combination of PRISMA-7, TUG and CDT. Additional clinical data and outcomes will be obtained from the electronic medical records of Landspítali. The postoperative outcomes measured will be 180-day mortality, surgical complications, 90-day readmission, delirium, non-home discharge and length of hospital stay.

Patients who screen positive on the CDT (≤ 2/3 points) and TUG (≥ 11 seconds) will be considered frail. Those who do not screen positive on both of these tests will be part of the control group (non-frail).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 70 years who present for preoperative work-up at the anesthesia department at Landspitali.
* Patients assigned to undergo intermediate/major surgery

Exclusion Criteria:

* Not undergoing planned surgery

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The study population will consist of all patients ≥70 years who present for preoperative assessment with an anesthesiologist at Landspitali before undergoing intermediate/major surgery, The National University Hospital of Iceland.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-21 (Estimated)

PRIMARY OUTCOMES:
Moderate and severe surgical complications (Clavien-Dindo ≥2) | Time frame: From the same day after surgery to postoperative day 30.
  Description: This outcome measures the incidence of adverse events after surgery and will be categorized based on the Clavien-Dindo classification grading system using the cut-off of ≥2; complications requiring pharmacological intervention (grade II), requiring additional procedures (grade III), life-threatening complications(grade IV) and a complication resulting in death (grade V).
90-day Readmission | From the day of surgery to postoperative day 90.
  Readmission to any hospital in Iceland where the patient is admitted to any inpatient department. Emergency department enrollment without admission will not be counted as readmission. A patient´s readmission on the same day of discharge is considered a single continuous admission, unless it is clear the reason for readmission is not related to the initial admission or surgery. In which case it would be considered a separate readmission.

SECONDARY OUTCOMES:
Length of hospital stay | From the day of primary surgery until discharge from the index hospitalization (same-day discharge counted as 0 days), assessed up to 180 days postoperatively.
  Length of the primary hospital stay after surgery, measured in days. Same-day discharge will be counted as 0, discharge on postoperative day 1 will be counted as 1, etc. A patient's readmission on the same day of discharge is considered a single continuous admission, unless the reason for readmission is clearly unrelated to the initial admission or surgery, in which case it will be considered a separate admission.
Postoperative delirium during primary hospitalization | From the day of surgery (postoperative day 0) until first documented postoperative delirium or discharge from the index hospitalization, whichever occurs first, assessed up to 180 days postoperatively.
  Any mention of postoperative delirium during the primary hospitalization in nursing/physician notes will be used to identify delirium.
Short-term mortality | Up to 1 year after the primary surgery
  Defined as the death of the patient after surgery
Non-home discharge | From the day of surgery (postoperative day 0) until discharge to a non-home destination or discharge from the primary hospitalization, whichever occurs first, assessed up to 180 days postoperatively.
  Non-home discharge will be identified as the postoperative hospital discharge to a nursing home or a rehabilitation center. Discharge to patient hotels will not be included. In addition, non-home discharge will not include patients who live in a nursing home prior to the surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Landspitali - The national university hospital in Iceland., Reykjavik, Hofudborgarsvaedid, Iceland

IPD SHARING:
Plan to Share IPD: No
The individual participant data collected during this study will not be shared due to confidentiality. Additionally, there is no formal plan for making these data publicly available at this time.

REFERENCES:
- [Background] Rabelo LG, Bjornsdottir A, Jonsdottir AB, Einarsson SG, Karason S, Sigurdsson MI. Frailty assessment tools and associated postoperative outcomes in older patients undergoing elective surgery: A prospective pilot study. Acta Anaesthesiol Scand. 2023 Feb;67(2):150-158. doi: 10.1111/aas.14162. Epub 2022 Nov 9. PMID 36307919